CLINICAL TRIAL: NCT01300221
Title: Real-time 3-Dimensional Echocardiography for Assessment of Cardiac Function and Congenital Heart Disease
Acronym: 3DE-CHD
Status: Withdrawn | Type: Observational
Why Stopped: Study did not receive IRB approval.
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Other Study IDs: H-16888
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Congenital Heart Disease
Keywords: Three dimension echocardiography; Congenital heart disease; Z-score
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Group 1: Subjects who are healthy normal children.
- Group 2: Subjects who have congenital heart disease.
- Group 3: Subjects who have sickle cell disease
- Group 4: Subjects who have Duchenne muscular dystrophy
- Group 5: Patients who have Marfan syndrome and other aortic disease

SUMMARY:
The propose of this study is to generate normative data of the tree-dimensional echocardiographic(3-DE) measurements for cardiac structure and function in a large cohort of normal infants, children,and adolescents. The investigators also sought to investigate the utility of 3-DE in evaluating infants, children and adolescents with congenital and acquired heart diseases.

DETAILED DESCRIPTION:
I. SPECIFIC AIMS

1. To measure and calculate Z Scores of cardiac structures and function using 3-DE in a large cohort of healthy infants, children, and adolescents.
2. To investigate the utility of 3-DE in infants, children and adolescents with congenital and acquired heart disease.

II. BACKGROUND AND SIGNIFICANCE

Congenital heart disease (CHD)is one of the most common congenital malformations and is associated with significant mortality and morbidity. Acquired heart diseases are also common and have significant impact on the health of the young. As the therapeutic strategies are evolving, reliable non-invasive methods to image the cardiovascular system and quantitatively assess cardiac function with accuracy and reproducibility are pivotal to define the natural history, to evaluate the results of intervention and to assess long-term outcome.Three-dimensional echocardiography (3-DE) has important clinical applications to CHD. Because of growth throughout childhood,interpretation of these measurements requires normalization of the dimensions of cardiac structures to the size of the body. This is commonly done by the calculation of Z scores for the measurement of interest. Currently available normative data in the medical literature are limited to one-dimensional and two-dimensional echocardiography measurements only.

In this study, we will generate normative data of the 3-DE measurements for cardiac structure and function in a large cohort of healthy infants, children,and adolescents. We will also investigate the utility of 3DE for assessing the cardiovascular structures and cardiac function for congenital and acquired heart disease.

III. DESIGN AND METHODS

A. Subjects:

A total of 800 study subjects will be enrolled in the study after approval by the Institutional Review Board. Echocardiography data will be prospectively collected. The subjects will be divided into 5 groups:

Group 1. (n=300) Patients with normal cardiac anatomy and function by echocardiography.

Group 2. (n=300) Patients with various congenital heart diseases.

Group 3. (n=100) Patients with sickle cell disease and at risk for ventricular remodeling and pulmonary hypertension.

Group 4. (n=50) Patients with Duchenne and muscular dystrophy at risk for ventricular remodeling and dysfunction.

Group 5. (n=50) Patients with Marfan syndrome or the aortic disease.

B. Procedure:

Before the study, heart rate and blood pressures will be obtained for each study subject. The subjects will be placed in a left recumbent position and ECG attached. After a complete conventional echocardiographic assessment of each subject, real-time 3-DE /Doppler study will be performed with 3-DE system. The 3-DE study will take about 30 minutes. After each study, all data will be saved and processed off line. Indication for the clinical echocardiogram will include cardiac murmur, syncope or chest pain but with a normal echocardiogram. Informed consent will be obtained from each patient and legal representatives after a full explanation of the procedure.

1. Conventional echocardiography All patients will undergo a complete 2- dimensional, color flow Doppler, and spectral Doppler examination. Examination will be performed using a commercially available ultrasound system (IE33 system, Philips, Andover, Mass). All measurements will be made offline using a computer workstation(Xcelera,Philips Medical Systems,Andover,MA). All measurements will be made according to American Society of Echocardiography protocol. For any given structure, measurement will be made if excellent and unambiguous views were available.
2. Transthoracic 3-DE The 3-DE/Doppler studies will be performed using the IE33 (Philips, Andover, MA,USA) ultrasound machine with X3-1 or X7-2 matrix-array transducers. The X7-2 matrix-array transducer is a new tool and particularly well suited for small children. The patient will be in a decubitus position. Image acquisition will be performed from an apical window with the LV as the region of interest based on international recommendations. To encompass the complete LV into the 3D dataset, a full volume scan will acquire in harmonic mode from four R-wave triggered subvolumes. This scan will carried out during an end-expiratory breath hold a few seconds when possible. The 3D dataset will be stored in a DICOM format on a CD-ROM and transferred to separate workstations for off-line data analysis.

C. Image off-line analysis

1. QLAB Semiautomated Border Detection Method:A semiautomated border detection biplane LV volume analysis was performed using off-line QLAB version 8.0 software (Philips). The LV end-diastolic volume (EDV) and end-systolic volume (ESV) (smallest LV volume) frames are identified.On both of these end-diastolic and end-systolic frames,five identification points are marked: the septal, lateral, anterior, and inferior mitral annulus and the apex (from either one of the views). Then the software automatically delineates the LV endocardial border and, by sequential analysis, creates a LV mathematical model or "cast" that represents the LV cavity.
2. TomTec Semiautomated Method:LV volume analysis will be performed off-line using TomTec 4D LV-Analysis software. TomTec requires triplane manual tracing of the endocardial border after which the software selects a fitting geometric model and the total LV endocardial border is automatically delineated with possible manual corrections. Based on the six initial contours, a spatiotemporal interpolation model (like a pulsating balloon) is created by rotational and temporal interpolation of these contours. According to the initial balloon, the algorithm starts to detect the endocardial border continuously in the entire 4D dataset (without large gaps due to interpolation), like deforming the balloon in the LV until it best fits the walls in each frame. Adjustments can be made manually after this step in oblique, sagittal, and coronal planes. Subsequently, a final reconstruction of the LV model and a time-volume curve are created. LV-EDV and LV-ESV are the largest and smallest volume, respectively, from this time-volume curve.

D. Data Analysis

All numerical values are expressed as mean +/- standard deviation. The real- time 3-DE measurements will be compared with other clinical data and measurements, such as cardiac catheterization or magnetic resonance imaging. Statistical significance will be defined as P<0.05. All statistical analyzes will be done using SAS for Windows version9.1 and Microsoft Excel (Microsoft Office 2007) for all analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosis that fits into Group 1 to 5 and who are willing to participate (consent/assent obtained)
* Do not meet the exclusion criteria (as follows).

Exclusion Criteria:

* Unwilling to participate or give consent.
* Clinically unstable.
* Unable to co-operate.
* Poor acoustic windows.

Ages: 1 Hour to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Group 1. (n=300) Subjects who are healthy normal children. Group 2. (n=300) Subjects who have congenital heart disease. Group 3. (n=100) Subjects who have sickle cell disease. Group 4. (n=50) Subjects who have Duchenne muscular dystrophy. Group 5. (n=50) Subjects who have Marfan syndrome and aortic disease.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shuping Ge, MD, Principal Investigator — Drexel University College of Medicine/St. Christopher's Hospital for Children
Locations (1):
- Drexel University College of Medicine/St. Christopher's Hospital for Children, Philadelphia, Pennsylvania, United States